CLINICAL TRIAL: NCT02796807
Title: Correlation Between SUV on 68Ga-HBED-CC-PSMA and Gleason Score in Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sir Mortimer B. Davis - Jewish General Hospital (Other)
Responsible Party: Principal Investigator, Stephan Probst, MD, Sir Mortimer B. Davis - Jewish General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 16-052
Record Dates: First submitted 2016-05-31; First posted 2016-06-13 (Estimated); Last update posted 2018-03-06 (Actual); Status verified 2018-03

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — gallium 68 PSMA-11

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 68Ga-HBED-CC-PSMA (DKFZ-11) PET/CT (Experimental)
  Interventions: Drug: 68Ga-HBED-CC-PSMA (DKFZ-11) PET/CT

INTERVENTIONS:
Drug: 68Ga-HBED-CC-PSMA (DKFZ-11) PET/CT

SUMMARY:
Prostate cancer is the second leading cause of cancer death in North American men older than 50 years. Prostate specific membrane antigen (PSMA) is a unique membrane bound glycoprotein, which is overexpressed manifold on prostate cancer cells and is well-characterized as an imaging biomarker of prostate cancer. Positron emission tomography / computer tomography (PET/CT) is a nuclear medicine procedure based on the measurement of positron emission from radiolabeled tracer molecules. 68Ga-HBED-CC-PSMA (DKFZ-11) (abbreviated 68Ga-PSMA) is a tracer for prostate cancer PET imaging. The strength of functional imaging methods is in distinguishing tissues according to metabolism rather than structure. Studies have shown that PET/CT imaging with 68Ga-PSMA can detect prostate cancer lesions with excellent contrast and a high detection rate even when the level of prostate specific antigen is low.

Study Objectives:

The objective of this study is to evaluate if the patient-wide SUVmax on 68Ga-PSMA PET/CT in locoregional and metastatic prostate cancer correlates with histopathologic Gleason score at initial biopsy. It is hypothesized that SUVmax will correlate positively with Gleason score. This is of interest because non-invasive risk stratification may be possible in the future.

This will be a single-site JGH-only open label study in which one (1) 68Ga-PSMA PET/CT will be performed on study participants. A PET/CT scan takes 2-3 hours.

ELIGIBILITY:
Inclusion Criteria:

* Resident of Canada
* Male sex
* Age 18 years or older
* Previous diagnosis of prostate cancer with Gleason Score available
* ECOG performance status 0 - 3, inclusive
* Able to understand and provide written informed consent
* Referred by a treating physician
* Able to tolerate the physical/logistical requirements of a PET/CT scan including lying supine for up to 45 minutes with the arms above the head and tolerating intravenous cannulation for injection of the study drug

Exclusion Criteria:

* Medically unstable patients (e.g. acute cardiac or respiratory distress or hypotensive, etc.)
* Patients who exceed the safe weight limit of the PET/CT bed (200 kg) or who cannot fit through the PET/CT bore (70 cm diameter)
* Patients who are claustrophobic

Ages: 18 Years to 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
SUVmax on 68Ga-PSMA PET/CT in locoregional and metastatic prostate cancer | Through study completion, one day

CONTACTS AND LOCATIONS:
Locations (1):
- Jewish General Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No